CLINICAL TRIAL: NCT07258602
Title: In-depth Interviews to Explore Patient and Partner/Caregiver Experiences, Unmet Needs, and Care Barriers in Patients With Implantable Cardioverter-defibrillators
Brief Title: In-depth Interviews of Patients With ICDs
Acronym: QoLICD-INSIGHT
Status: Enrolling by invitation | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S71109
Record Dates: First submitted 2025-09-24; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Implantable Cardioverter Defibrillator (ICD)
Keywords: quality of life; implantable cardioverter defibrillator (ICD)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: semi-structured interview — Patients with an ICD and partner/caregivers will be invited for semi-structured interviews interviews to explore how ICD patients and their partners/caregivers interpret and navigate these challenges in their own words. Interviews provide a richer understanding of personal experiences, unmet needs, and barriers to care that are not easily measurable through questionnaires alone. Including both patients and their partners offers insight into relational dynamics and caregiving perspectives.

SUMMARY:
Although ICDs are effective in preventing sudden cardiac death, they can also profoundly affect patients' and partner/caregivers' emotional well-being, social relationships, and daily functioning. Previous phases of the QoL-ICD project used patient-reported outcome measures (PROMs) and support group discussions to identify key domains affecting quality of life: patient education, physical health, psychological and social well-being, and end-of-life awareness. However, these methods have limitations in capturing the full depth and context of lived experience.

To complement and expand on these findings, this study uses in-depth, semi-structured interviews to explore how ICD patients and their partners interpret and navigate these challenges in their own words. Interviews provide a richer understanding of personal experiences, unmet needs, and barriers to care that are not easily measurable through questionnaires alone. Including both patients and their partners offers insight into relational dynamics and caregiving perspectives.

The primary objective of this study is to explore the lived experiences of ICD patients and their partners across four key domains:

* Patient education and information provision
* Physical health and activity
* Psychological and social well-being
* End-of-life considerations

DETAILED DESCRIPTION:
The investigators will ensure purposive sampling across key demographic and clinical variables which are available after a participant has expressed interest in the trial, with a minimum of 15 participants with ICD per subgroup (e.g., sex, age category, underlying cardiac condition). Data collection will continue until thematic saturation is reached within the overall cohort, followed by at least 5 additional interviews to confirm stability of themes. Subgroup representation is intended to capture relevant variation in lived experience and ensure applicability of findings across the ICD population. There is no subgroup analysis scheduled for partners as this cohort is considered secondary.

Predefined subgroups of interest:

* Sex
* Age: <35 years; 35 to 65 years; and > 65 years
* Underlying cardiac condition: congenital heart disease, hypertrophic cardiomyopathy, primary arrhythmia syndromes, Ischemic cardiomyopathy, Non-ischemic cardiomyopathy
* ICD shock history: appropriate ICD shock; inappropriate ICD shock; none
* Time since implantation: cut-off at 2 years
* ICD indication: primary vs secondary prevention
* Device type: single/dual/S-ICD vs cardiac resynchronization therapy

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years) with an implanted ICD for either primary or secondary prevention of sudden cardiac death.
* At least 3 months have passed since ICD implantation.
* Sufficient cognitive ability and fluency in Dutch to provide informed consent and actively participate in the interview.
* Willing and able to participate in a one-time, individual in-depth interview of 30 to 60 minutes.

Exclusion Criteria:

* Current active severe psychiatric disorder or cognitive impairment that would interfere with meaningful participation as based on the medical history..
* Inability to provide informed consent due to legal, cognitive, or communicative limitations.
* Medical instability or terminal illness that, in the opinion of the treating physician or research team, precludes participation.
* Participation in another interventional trial that may influence psychological or behavioral outcomes relevant to this study.
* Participation in the QoL-ICD II trial with longitudinal QoL assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with any type of implantable cardioverter-defibrillator followed at UZ Leuven and their partners or primary caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Thematic saturation across interviews of the 4 predefined domains | 1 year
  This qualitative study has descriptive and thematic endpoints, not statistical. The primary endpoint is defined as thematic saturation across interviews regarding 4 predefined domains: patient education and information provision, physical health and activity, psychological and social well-being, and end-of-life considerations. Thematic saturation indicates that the data collected sufficiently captures the full range of relevant experiences, perspectives, and needs of ICD patients and their partners. To track thematic saturation a saturation grid and theme tracking table will be used.
  A saturation grid tracks the appearance of themes and documents: (1) themes present in each interview; (2) when new themes emerge; (3) when previously identified themes are reinforced. Theme tracking tables summarize the progress by coding the number of new themes. Thematic saturation is reached when 5 consecutive interviews fail to produce any new themes after a minimum of 15 interviews per subgroup.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided